CLINICAL TRIAL: NCT03359044
Title: Bronchoscopy Anesthesia and Neuropsychological Assessment in Children (BANACH) Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2017-03-208
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2017-10

CONDITIONS: Pneumonia; Atelectasis; Cough
Keywords: Fiberoptic bronchoscopy; Neuropsychological Development; general anesthesia
MeSH Terms: conditions — Pneumonia; Pulmonary Atelectasis; Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sedation + topical anesthesia: midazolam 0.1～0.2 mg/kg for sedation, 2%lidocaine for topical anesthesia
- General anesthesia+ topical anesthesia: propofol 4～5mg/kg、Remifentanil2～3μg/kg for induction ,insert Laryngeal Mask Airway(LMA) , 2%lidocaine for topical anesthesia

SUMMARY:
Fiberoptic bronchoscopy plays a very important role in the diagnosis and treatment of respiratory diseases in children.In China,this procedure is mainly performed under two different anesthesia methods：sedation and general anesthesia(GA) . Which is better ? there are still a lot of controversies . Several early retrospective studies suggest that, in addition to the possible increase in costs, general anesthesia in intraoperative complications, postoperative recovery and other aspects did not bring significant improvement. But clinically we observed that children under sedation often can not cooperate, they often shows anxiety,restless,crying,and so on, under these situation, some restraint measures may be used, which may have an impact on the child's neuropsychological development. Therefore ,we design this study ,aiming to compare the influence between sedation and general anesthesia (GA) on children 's neuropsychological development.

ELIGIBILITY:
Inclusion Criteria:

* Age 4-10 years
* American society of anesthesiologists(ASA) gradeⅠ～Ⅱ
* Plan to accept fiberoptic bronchoscopy treatment
* lives in the city where the research unit is located
* signed informed consent

Exclusion Criteria:

* preterm infants less than 28 weeks of gestational age or preoperative screening found that development, cognitive or behavioral abnormalities
* known congenital malformations may have a potential impact on the development of children's neuropsychological function
* known to have central nervous system disorders or meet the diagnostic criteria of Diagnostic and Statistical Manual(DSM) mental illness
* children with contraindications to intravenous general anesthesia

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: (1)Age 4-10Years;(2)ASAⅠ～Ⅱ;(3)Plan to accept fiberoptic bronchoscopy treatment;(4) lives in the city where the research unit is located;(5)signed informed consent
Sampling Method: Non-Probability Sample
Enrollment: 290 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
The detection rate of abnormal behavior in both groups | Three years after operation
  Using the Achenbach Child Behavior Checklist(CBCL)for Parents.The CBCL is a widely used parent report questionnaire identifying behavioural and emotional problems in children. The CBCL is administered in interview format and respondents are asked to rate 112 problem items as 0 for "not true of the child," 1 for "somewhat or sometimes true of the child," and 2 for "very true or often true of the child", based on the past two months. The raw scores from the 112 items are then compared with age- and gender-matched controls from the standardization sample, and standard scores are then derived with a mean of 50 and a standard deviation of 10. Worst value is 80; best value is 30.

SECONDARY OUTCOMES:
Full Scale Intelligence Quotient (FSIQ) Score of the Wechsler Intelligence Scale for Children (WISC)-IV | Three years after operation
  The WISC-IV is designed for children 6 years 0 months to 16 years 11 months. This study used the Full Scale IQ, which ranges from 45 to 155 with a mean of 100 and standard deviation of 15. Higher scores indicate stronger cognitive function. Scores between 90 and 110 are considered to be within the range of average IQ